CLINICAL TRIAL: NCT06251245
Title: The Effects of Different Methods Used in Oral Drug Administration on Fear in Children with Fever
Brief Title: The Effects of Different Methods Used in Pediatric Oral Drug Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Principal Investigator, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2023/10
Record Dates: First submitted 2024-02-02; First posted 2024-02-09 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Children, Only; Fear
Keywords: oral medication administration; fear; children; pediatric nursing
MeSH Terms: interventions — spoon protein, Drosophila

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Oral Injector) (Experimental): Children who use oral injectors to give oral medication will constitute the experimental group.
  Interventions: Procedure: Oral Injector
- Control group (Spoon) (Other): Children who use spoons to give oral medication will constitute the control group.
  Interventions: Procedure: Spoon

INTERVENTIONS:
Procedure: Oral Injector — * Admission of a child with fever to the pediatric inpatient ward
  * Obtaining parental consent
  * Completing the patient identification data collection form
  * Obtaining the child's consent
  * Applying the "Child Fear Scale" to the child
  * Measuring the child's pulse and SpO2
  * Applying the "Child Fear Scale" to the parent
  * Explaining the procedure using the educational therapeutic play method before oral medication administration
  * Administering the "Child Fear Scale" to the child and parent before oral medication administration
  * Measurement of the child's pulse and SpO2
  * • Experimental Group (Giving the medicine orally to the child with an Oral Injector)
  * Application of the "Child Fear Scale" to the child and parent after oral medication administration
  * Measurement of the child's pulse and SpO2
  Arms: Experimental Group (Oral Injector)
Procedure: Spoon — * Admission of a child with fever to the pediatric inpatient ward
  * Obtaining parental consent
  * Completing the patient identification data collection form
  * Obtaining the child's consent
  * Applying the "Child Fear Scale" to the child
  * Measuring the child's pulse and SpO2
  * Applying the "Child Fear Scale" to the parent
  * Explaining the procedure using the educational therapeutic play method before oral medication administration
  * Administering the "Child Fear Scale" to the child and parent before oral medication administration
  * Measurement of the child's pulse and SpO2
  * Control Group (Giving the medicine orally to the child with an oral medication spoon)
  * Application of the "Child Fear Scale" to the child and parent after oral medication administration
  * Measurement of the child's pulse and SpO2
  Arms: Control group (Spoon)

SUMMARY:
The aim of this study is to determine the effect of the use of spoons and oral injectors on the level of fear in children with fever in oral medication administration.

DETAILED DESCRIPTION:
Fever is known as a defense mechanism of the body; Increased body temperature in children is one of the symptoms that frighten parents and is among the most common reasons for hospitalization. Pharmacological agents such as paracetamol and ibuprofen are often used in fever management, and if possible, oral administration of the suspension form of the drugs is preferred to reduce invasive practices. However, reasons such as children not liking the taste of the medicine, rejecting the medicine, or spitting or vomiting may cause difficulties in administering the medicine orally. More than one different method is used to administer these drugs, depending on the patient's age, general condition and compliance with the treatment. These; They can be listed as spoon, oral injector, medicine glass. As a result of the examination of the drug administration materials, it was stated that children are fear of the injector when the drugs are given with a injector, they may aspirate, and they do not have appropriate equipment to administer the drug. It is important for nurses to understand children's fears and their causes, to develop interventions to reduce fear, and to minimize possible traumatic effects during the hospitilization process.

In this study, the sample will be divided into two groups: experimental and control, and oral antipyretic medicine will be given by two different methods. An oral injector will be used in the experimental group and an oral medicine spoon will be used in the control group.

Hypotheses of the Study:

H0: There is no significant difference in the effect of the use of spoons and oral injectors in oral medication administration in children on the level of fear in children and parents.

H1: There is a significant difference in the fear level of using spoons and oral injectors in oral medication administration in children.

H2: There is a significant difference in the parents' fear level of using spoons and oral injectors in oral medication administration in children.

H3: There is a significant difference in the heart rate and oxygen saturation of children using spoons and oral injectors for oral medication administration.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-6 and their parents,
* Children with fever,
* Children who have been ordered to take oral medication for fever in their treatment,
* Able to express himself cognitively,
* Able to speak and understand Turkish

Exclusion Criteria:

* Children who have a disease that may prevent them from expressing their fear
* It is time for the child to sleep at the time of medication administration.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Change in the child's fear level | at the time of admission to the hospital, immediately before oral medication administration, immediately after medication administration. The change in these time intervals will be assessed
  Child Fear Scale is used to measure the level of fear in children. This scale consists of five different facial expressions ranging from 0 = this face is not afraid at all to 4 = the most fear possible. The child and the parents are asked to look at these faces and choose the most appropriate expression to describe their fear. It is used in both children and parents to evaluate fear before and during the procedure
Change in parent's fear level | at the time of admission to the hospital, immediately before oral medication administration, immediately after medication administration. The change in these time intervals will be assessed
  Child Fear Scale is used to measure the level of fear in children. This scale consists of five different facial expressions ranging from 0 = this face is not afraid at all to 4 = the most fear possible. The child and the parents are asked to look at these faces and choose the most appropriate expression to describe their fear. It is used in both children and parents to evaluate fear before and during the procedure
Change in child's heart rate | at the time of admission to the hospital, immediately before oral medication administration, immediately after medication administration. The change in these time intervals will be assessed
  This outcome will be considered as one of the vital signs. Heart rate measurement will be evaluated via monitor.
Change in child's oxygen saturation | at the time of admission to the hospital, immediately before oral medication administration, immediately after medication administration. The change in these time intervals will be assessed
  This outcome obtained with patient monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Health Group, Ataşehir Hospital, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akram G, Mullen AB. Paediatric nurses' knowledge and practice of mixing medication into foodstuff. Int J Pharm Pract. 2012 Jun;20(3):191-8. doi: 10.1111/j.2042-7174.2011.00179.x. Epub 2011 Nov 9. PMID 22554162
- [Background] Alessandrini E, Walsh J, Salunke S. Usability of administration devices for oral and respiratory medicines: Views from a UK primary school. Eur J Pharm Biopharm. 2022 Sep;178:150-158. doi: 10.1016/j.ejpb.2022.08.006. Epub 2022 Aug 17. PMID 35987466
- [Background] Chiappini E, Venturini E, Remaschi G, Principi N, Longhi R, Tovo PA, Becherucci P, Bonsignori F, Esposito S, Festini F, Galli L, Lucchesi B, Mugelli A, Marseglia GL, de Martino M; Italian Pediatric Society Panel for the Management of Fever in Children. 2016 Update of the Italian Pediatric Society Guidelines for Management of Fever in Children. J Pediatr. 2017 Jan;180:177-183.e1. doi: 10.1016/j.jpeds.2016.09.043. Epub 2016 Oct 31. PMID 27810155
- [Background] Talegaonkar S, Chitlangia A, Pradhan V, More S, Salunke S. Uncovering caregiver concerns: 5 key issues that still remain unresolved in administration of oral medicines for children in India. Eur J Pharm Biopharm. 2023 Jun;187:166-174. doi: 10.1016/j.ejpb.2023.03.009. Epub 2023 Mar 23. PMID 36965592
- [Background] Turgut MA, Turkmen AS. The effect of lighted toy on reducing pain and fear during blood collection in children between 3 and 6 years: A randomized control trial. J Pediatr Nurs. 2023 May-Jun;70:111-116. doi: 10.1016/j.pedn.2023.02.009. Epub 2023 Mar 9. PMID 36905910